CLINICAL TRIAL: NCT01739296
Title: Lateral Wedge Insole With Subtalar Strapping for Knee Osteoarthritis: a Randomized Clinical Trial
Brief Title: Lateral Wedge Insole With Subtalar Strapping for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 839/2011
Record Dates: First submitted 2012-11-22; First posted 2012-12-03 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; osteoarthritis, knee; foot orthoses; orthotic insoles
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wedge (Experimental): Lateral wedge insole with subtalar strapping Use of lateral wedge insoles with subtalar strapping for 5 to 10 hours daily
  Interventions: Other: Lateral wedge insole with subtalar strapping
- Neutral (Sham Comparator): Neutral insole with subtalar strapping (sham) Use of neutral insoles with subtalar strapping for 5 to 10 hours daily
  Interventions: Other: Neutral insole with subtalar strapping (sham)

INTERVENTIONS:
Other: Neutral insole with subtalar strapping (sham) — Neutral insole with subtalar strapping (sham)
  Other Names: Neutral
  Arms: Neutral
Other: Lateral wedge insole with subtalar strapping — Lateral wedge insole with subtalar strapping
  Other Names: Wedge
  Arms: Wedge

SUMMARY:
This is a clinical study to evaluate the efficacy of a lateral wedge insole with subtalar strapping in knee osteoarthritis treatment.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the efficacy of a lateral wedge insole with subtalar strapping in knee osteoarthritis treatment. Fifty-eight patients with knee osteoarthritis were randomized to use either a lateral wedge or a neutral insole. VAS, Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and Lequesne questionnaires were applied at baseline, and weeks two, eight, and 24.

ELIGIBILITY:
Inclusion Criteria:

* Meet the American College of Rheumatology criteria for knee Osteoarthritis
* Varus malalignment of the knee
* Absence of previous fracture on the index knee
* Absence of previous surgery on the index knee
* Absence of Rheumatoid Arthritis
* No Intra-articular injection on the index knee in the past 6 months
* Receiving usual care for Osteoarthritis for at least 6 months
* Be able to understand and agree with the informed consent

Exclusion Criteria:

* Undergo surgery during the study
* Undergo Intra-articular injection during the study
* Develop articular infection of the index joint during the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Symptoms | 24 weeks
  Evaluation of patient's symptoms using WOMAC (western ontario and mcmaster universities osteoarthritis index), VAS (visual analogic scale of pain) and Lequesne questionaires

SECONDARY OUTCOMES:
Ankle pain | 24 weeks
  Number of patients that reported ankle pain related to the use of the insole as a measure of tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo C Campos, MD, Principal Investigator — FMUSP
Locations (1):
- Instituto de Ortopedia e Traumatologia HC-FMUSP, São Paulo, São Paulo, Brazil

REFERENCES:
- See also: Brazilian Orthopaedics Association — http://sbot.org.br
- See also: Orthopaedics and Traumatology Institute website — http://iothcfmusp.com.br
- See also: University of São Paulo website — http://fmusp.org.br
- See also: Brazilian Knee Surgery Association website — http://sbcj.org.br